CLINICAL TRIAL: NCT06630780
Title: A Prospective Phase II Clinical Trial on the Reduction of Postoperative Radiotherapy in Head and Neck Squamous Cell Carcinoma
Brief Title: Reduction of Postoperative Radiotherapy in Head and Neck Squamous Cell Carcinoma
Acronym: REPORT-HNSCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chen Chunyan, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-FXY-224
Record Dates: First submitted 2024-09-17; First posted 2024-10-08 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC)
Keywords: HNSCC; Post-radical surgery; Adjuvant Radiotherapy; Radiation dose reduction; Quality of life
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: Phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Trial Group (Experimental): All patients received intensity-modulated conformal radiotherapy (IMRT). To ensure study quality, all IMRT plans were reviewed by the research team at Sun Yat-sen University Cancer Center. The delineation principles for the radiotherapy target volume of the primary tumor bed and normal tissues followed the consensus guidelines.
  (1) Tumor bed (CTVtb): It was delineated based on the tumor extent shown in laryngoscopy, enhanced CT/MRI, or PET CT before induction therapy49. For patients with significant anatomical changes due to tumor regression, the CTVtb was adjusted, taking into account the patient's anatomy after induction chemotherapy and the initial state of the tumor; if a cavity appeared due to tumor regression, it was adjusted according to natural anatomical boundaries.(2) High-risk clinical target volume (CTV1): CTVtb plus a 5-10mm margin, with a prescribed dose of at least 60Gy in 30 fractions.
  (3) Low-risk clinical target volume (CTV2): CTV1 plus a 5-10mm margin. For hypo
  Interventions: Radiation: Head and Neck Cancers

INTERVENTIONS:
Radiation: Head and Neck Cancers — All patients received intensity-modulated conformal radiotherapy (IMRT). To ensure study quality, all IMRT plans were reviewed by the research team at Sun Yat-sen University Cancer Center. The delineation principles for the radiotherapy target volume of the primary tumor bed and normal tissues followed the consensus guidelines.

SUMMARY:
To explore the control rate and quality of life of participants with late head and neck squamous cell carcinoma who have obtained postoperative pCR after cervical lymph node surgery with neoadjuvant chemotherapy combined with immunotherapy, and the cervical lymph node removal prophylactic irradiation ENI in the low-risk area.

DETAILED DESCRIPTION:
In order to understand whether it can better protect normal tissues such as pharyngeal constriction muscles, thyroid, parotid glands, and submandibular glands without affecting the efficacy of tumors, and reduce the negative impact of radiotherapy on immunotherapy, the investigators plan to conduct a prospective phase II study to explore the control rate and quality of life of patients with late head and neck squamous cell carcinoma who have obtained postoperative pCR after cervical lymph node surgery with neoadjuvant chemotherapy combined with immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative pathologically confirmed initial treatment of head and neck squamous cell carcinoma
* Receive neoadjuvant chemotherapy combined with PD-1 monoclonal antibody immunotherapy, and meet one of the following conditions: Preoperative clinical stage was T3-T4 or N2-N3 (AJCC 8th edition). Patients with oral cancer/oropharyngeal cancer had positive lymph nodes in the IV/V region with imaging diagnosis or biopsy confirmation before surgery. HPV/ P16-positive oropharyngeal cancer patients with clinical lymph node invasion (ENE), one positive cervical lymph node > 3cm or multiple positive cervical lymph nodes before surgery
* The pathology of at least one cervical lymph node was determined by pCR；
* Karnofsky's physical status score ≥70 points；
* Age: 18 ~ 70 years old；
* Laboratory examination results within 1 week before enrollment met the following conditions: neutrophils (ANC) ≥1.5×109/L, platelets (PLT) ≥ 75×109/L
* Patients participate voluntarily and sign informed consent forms.

Exclusion Criteria:

* Previous head and neck radiation treatment
* Severe complications；
* Pregnant or lactating women
* Who were deemed unsuitable for inclusion by the researchers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year region-free recurrence survival (RRFS) | 2-year
  Time to confirmed diagnosis of documented recurrence of cervical lymph nodes or death from any cause

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2-year
  Defined as documented treatment progression or death from any cause.
Distant metastasis-free survival (DMFS) | 2-year
  Defined as documented distant metastases or death from any cause
Overall survival (OS) | 2-year
  Defined as a documented death due to any cause or last follow-up; regional recurrence pattern; and acute and late toxicity.
Local recurrence-free survival (LRFS) | 2-year
  Defined as documented primary tumor recurrence or death from any cause
Acute and Late Radiation Injuries | Day 1 of radiotherapy to 2 years post-treatment
  The acute radiation toxicity was assessed using the CTCAE 5.0 version, while the RTOG and EORTC late radiation toxicity scales were used to evaluate late toxicity.
Quality of life assessment | Baseline, during radiotherapy, at the end of radiotherapy, 3 months after the end of radiotherapy, 6 months after the end of radiotherapy, and thereafter according to routine follow-up until 2 years.
  The Quality of Life (QoL) was assessed at baseline and during follow-up using the European Organization for the Head and Neck Cancer Module (QLQ-H&N35) version 1.0.
Quality of life assessment | Baseline, during radiotherapy, at the end of radiotherapy, 3 months after the end of radiotherapy, 6 months after the end of radiotherapy, and thereafter according to routine follow-up until 2 years.
  The Quality of Life (QoL) was assessed at baseline and during follow-up using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30).

CONTACTS AND LOCATIONS:
Overall Officials: Liu-Wei Tang, Study Director — The Ethics Committee of the Center for Cancer Prevention and Treatment, Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Data supporting this study's findings are available from the PI (Chun-Yan Chen) upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Commencing from the publication date of papers related to this study, with no end date.
Access Criteria: Data will be collected using a case record form (CRF). The PI will securely maintain all trial records, CRFs, and study-related documents for ten years in the study office before archiving them in the Medical Records section. Access will be provided to the PI, CIs, and IEC with the appropriate permissions. The PI will also be responsible for overseeing communication with the IEC and DSMU to ensure ethical oversight and participant safety.
URL: https://www.researchdata.org.cn/